CLINICAL TRIAL: NCT03598166
Title: Assessing the Effect of Offering a Blood-based Colorectal Cancer Screening Test on Screening Adherence and Colonoscopy Completion in Patients Who Have Refused Colonoscopy and FIT
Brief Title: Assessing the Effect of a Blood-based Colorectal Cancer Screening Test on Screening Adherence and Colonoscopy Completion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter S. Liang, MD MPH (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Peter S. Liang, MD MPH, Staff Physician, VA New York Harbor Healthcare System
Organization: VA New York Harbor Healthcare System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MIRB 01683
Record Dates: First submitted 2018-07-02; First posted 2018-07-26 (Actual); Results first posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer screening; septin 9
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized 1:1 to the intervention or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): Patients will receive a letter noting that they are not up-to-date on screening and encouraging them to contact a study number if they choose to screen with colonoscopy or FIT. Patients who call will speak to a research assistant who is trained in patient navigation and can facilitate referrals for colonoscopy or FIT. Patients will receive a follow-up telephone call that reiterates information in the letter.
  Patients will also be asked to complete a questionnaire about their beliefs and attitudes regarding CRC screening. The questionnaire will be mailed with the invitation letter and will also be administered over the telephone by the research assistant.
- Septin9 (Experimental): Patients will receive a letter noting that they are not up-to-date on screening and encouraging them to contact a study number if they choose to screen with colonoscopy or FIT. Letters will also include an option to participate in the blood test, with instructions to call the study number to schedule the blood draw. This option will not appear in the letters sent to the control group. Patients will also receive a follow-up telephone call and a questionnaire.
  Participants who choose to the blood test (Septin9) will undergo phlebotomy. The blood sample will be run by an off-site commercial laboratory. The study team will notify patients and their primary care physicians of blood test results and will facilitate a colonoscopy referral for those with positive tests.
  Interventions: Diagnostic Test: Septin9

INTERVENTIONS:
Diagnostic Test: Septin9 — Septin9 is a FDA-approved blood test for colorectal cancer screening
  Other Names: Epi proColon; Epigenomics
  Arms: Septin9

SUMMARY:
Objectives:

Colonoscopy and stool-based testing are the two predominant colorectal cancer (CRC) screening tests used in the US, and both reduce colorectal cancer mortality. However, only 62% of Americans are up to date with screening, partly because many individuals find these two tests inconvenient or unacceptable for a variety of reasons. There is an unmet need for a non-invasive test that does not require bowel preparation or handling stool, and the Septin9 DNA blood test may be an alternative for those individuals who would otherwise remain unscreened.

Aims:

Aim 1: To measure screening uptake with a blood test in screen-resistant patients who have declined both colonoscopy and fecal immunochemical testing (FIT) at the Manhattan VA Medical Center

* Sub-Aim 1a: To assess the proportion of those with a positive blood-based screening test who undergo diagnostic colonoscopy
* Sub-Aim 1b: To describe the endoscopic findings on diagnostic colonoscopy

Aim 2: To survey screen-resistant patients to understand their beliefs and attitudes about colorectal cancer screening and testing options

We hypothesize that a substantial proportion of patients who have refused colonoscopy and FIT will accept the blood test. We hypothesize this will be driven by the convenience of the blood test.

Methods:

This will be randomized controlled trial of individuals who have refused colonoscopy and FIT within past 6 months. Eligible patients will be randomized 1:1 to the intervention or control group. Both groups will be invited to participate in navigated colonoscopy or FIT by letter and telephone call. The intervention group will also be invited to participate in the blood test if they refuse colonoscopy and FIT. We will enroll 180 participants in each group (total n=360).

DETAILED DESCRIPTION:
The proposed study is a randomized controlled trial that will 1) assess the uptake of a CRC screening blood test among patients who have declined both colonoscopy and FIT in the previous 6 months, including diagnostic evaluation of positive results and 2) survey patients about their beliefs and attitudes regarding CRC screening and testing options. All participants will be primary care patients at the Manhattan VA Medical Center. Based on a recent internal audit, there were 1502 patients who had at least one primary care visit from August 2016 through August 2017 and were not up to date with CRC screening. Up-to-date CRC screening is defined as either 1) a colonoscopy within the past 10 years or 2) FIT within the past year. We will perform an updated CRC screening audit at the beginning of the study to obtain the entire pool of eligible patients who are not up to date with screening. Eligible patients will then be randomized 1:1 to either an intervention group or a control group. All patients will receive a letter noting that they are not up-to-date on screening and encouraging them to contact a study number if they choose to screen with colonoscopy or FIT. Patients who call will speak to a research assistant who is trained in patient navigation and can facilitate referrals for colonoscopy or FIT. Following the sequential testing approach, letters addressed to the intervention group will also include an option to participate in the blood test, with instructions to call the study number to schedule the blood draw. In addition to the letter, both groups will also receive a follow-up telephone call that reiterates information in the letter. The research assistant will make and receive all calls using a standard script. All patients will also be asked to complete a survey about their beliefs and attitudes regarding CRC screening. The survey will be mailed with the invitation letter and will also be administered over the telephone by the research assistant. The study team will notify patients and their primary care physicians of blood test results and will facilitate a colonoscopy referral for those with positive tests. Primary care physicians will not be asked to notify the patients or make the colonoscopy referral because most will not have adequate knowledge of the Septin9 test to provide appropriate patient education.

Participants who are randomized to the blood test arm will undergo phlebotomy, which will be performed by the study research assistant. The blood sample will be temporarily stored on-site and then transported to an off-site commercial laboratory (Lenco Diagnostic Laboratory, Brooklyn, NY) to run the assay.

Clinical outcomes for both the intervention and control group participants will be measured as a secondary outcome. This includes timing and result of a screening colonoscopy or FIT for individuals in the controls group as well as diagnostic colonoscopy for participants who had a positive blood test.

ELIGIBILITY:
Inclusion Criteria:

* not up-to-date with colorectal cancer screening, defined as a colonoscopy in the past 10 years, a stool test (FOBT/FIT) in the past year, or a flexible sigmoidoscopy in the past 5 years.
* Declined colorectal cancer screening (both colonoscopy and FIT) in the previous 6 months, which must be documented in the electronic health record

Exclusion Criteria:

* Personal history of colonic adenomas (including sessile serrated adenomas), proximal hyperplastic polyps, CRC, inflammatory bowel disease, or hereditary gastrointestinal cancer syndrome
* First degree relative with CRC diagnosed at <60 years of age; family history of hereditary gastrointestinal cancer syndromes.
* Vulnerable populations
* Adult unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VA New York Harbor Health Care System, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liang PS, Zaman A, Kaminsky A, Cui Y, Castillo G, Tenner CT, Sherman SE, Dominitz JA. Blood Test Increases Colorectal Cancer Screening in Persons Who Declined Colonoscopy and Fecal Immunochemical Test: A Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2023 Oct;21(11):2951-2957.e2. doi: 10.1016/j.cgh.2023.03.036. Epub 2023 Apr 8. PMID 37037262

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The target enrollment specified in the protocol is 360 participants. Actual enrollment was 359 participants.
Groups:
- Septin9: Patients will receive a letter noting that they are not up-to-date on screening and encouraging them to contact a study number if they choose to screen with colonoscopy or FIT. Letters will also include an option to participate in the blood test, with instructions to call the study number to schedule the blood draw. This option will not appear in the letters sent to the control group. Patients will also receive a follow-up telephone call and a questionnaire.
  Participants who choose to the blood test (Septin9) will undergo phlebotomy. The blood sample will be run by an off-site commercial laboratory. The study team will notify patients and their primary care physicians of blood test results and will facilitate a colonoscopy referral for those with positive tests.
  Septin9: Septin9 is a FDA-approved blood test for colorectal cancer screening
Period: Overall Study
Arm/Group | Control | Septin9
Started | 178 | 181
Completed | 178 | 181
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Individuals who are eligible for colorectal cancer screening and have previously declined colonoscopy and FIT.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Septin9 | Total
Number analyzed (Participants) | 178 | 181 | 359
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 76 | 87 | 163
  >=65 years | 102 | 94 | 196
Age, Continuous [Median (Full Range); unit: Years] | 67 [50 to 75] | 66 [50 to 75] | 66 [50 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 171 | 172 | 343
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 29 | 55
  Not Hispanic or Latino | 151 | 147 | 298
  Unknown or Not Reported | 1 | 5 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The analysis population is excluding Hispanics in this total, as it was already recorded in a different section. This is why the total is less than the original total.
  Participants
    number analyzed (Participants) | 152 | 152 | 304
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 3 | 2 | 5
    Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
    Black or African American | 70 | 77 | 147
    White | 68 | 62 | 130
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 178 | 181 | 359

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Undergo Screening Within 6 Months of Outreach
Description: Percentage of participants who undergo screening in the intervention group vs. control group, measured 6 months after the initial letter was sent
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Septin9
Number analyzed (Participants) | 178 | 181
Participants | 17 | 31

2. Secondary Outcome: Percentage of Participants Completing Screening Strategy
Description: Complete screening in both groups, which is defined as completion of the entire screening strategy. For colonoscopy, this requires cecal intubation and an adequate bowel preparation. For individuals who took Septin9 and FIT, positive results must be followed by a colonoscopy with cecal intubation and adequate bowel preparation.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Septin9
Number analyzed (Participants) | 178 | 181
Participants | 16 | 27

3. Secondary Outcome: Percentage of Participants With Colonoscopy Follow-up in Intervention Group
Description: Among individuals in the intervention group who had a positive blood test, proportion who completed a follow-up colonoscopy within 6 months.
Time Frame: 6 months (after positive FIT)
Population: The overall number of participants analyzed corresponds to the number of participants with a positive FIT.
Measure: Count of Participants; unit: Participants
Arm/Group | Septin9
Number analyzed (Participants) | 2
Participants | 1

4. Secondary Outcome: Self-reported Willingness to Take Blood Test for Colorectal Cancer Screening on Questionnaire
Description: Percentage of both groups who answered that they would be willing to take a blood test for colorectal cancer screening
Time Frame: 1 day (assessed using baseline survey)
Population: The same survey was sent to all participants. The planned analysis was to include all participants who returned the survey, rather than stratified by arm.
Measure: Count of Participants; unit: Participants
Groups:
- Surveys/Questionnaires Mailed: The survey was sent out to both control and intervention patients and all surveys contained the same questions. It investigated patients' perspectives on colonoscopy and FIT in order to understand barriers to screening. The survey also assessed whether these patients would be amenable to a blood-based CRC screening test.
Arm/Group | Surveys/Questionnaires Mailed
Number analyzed (Participants) | 76
Participants | 65

5. Secondary Outcome: Self-reported Most Common Advantages of Blood Test on Questionnaire
Description: The most commonly cited advantages of a blood test compared to colonoscopy and stool test in both groups
Time Frame: 1 day (assessed using baseline survey)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- Convenience: Patients are willing to go through a blood test for colorectal cancer screening due to the convenience of taking a blood test.
- No Special Preperation: Patients are willing to take blood tests for colorectal cancer screening due to a lack of extra preparation for a blood test.
- Accustomed to Blood Tests: Patients are willing to do a blood test for colorectal cancer screening because they feel accustomed to blood draw tests.
Arm/Group | Convenience | No Special Preperation | Accustomed to Blood Tests
Number analyzed (Participants) | 76 | 76 | 61
Participants | 46 | 31 | 24

6. Secondary Outcome: Self-reported Most Common Reasons for Refusing Blood Test on Questionnaire in Intervention Group
Description: The most commonly cited reasons for not taking the blood test in the intervention group.
Time Frame: 1 day (assessed using baseline survey)
Population: The overall number of participants who indicated that they would refuse a blood test on the questionnaire.
Measure: Count of Participants; unit: Participants
Groups:
- Not as Accurate as FIT: Patients who declined blood draws for colorectal cancer do not believe it is as accurate as the FIT test.
- Uncomfortable With Blood Draws: Patients who declined blood draws for colorectal cancer screening state they are uncomfortable with blood draws.
Arm/Group | Not as Accurate as FIT | Uncomfortable With Blood Draws
Number analyzed (Participants) | 9 | 9
Participants | 4 | 3

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Control | Septin9
All-Cause Mortality (participants affected / at risk) | 3/178 | 2/181
Serious Adverse Events (participants affected / at risk) | 0/178 | 0/181
Other Adverse Events (participants affected / at risk) | 0/178 | 0/181

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT03598166/Prot_SAP_001.pdf